CLINICAL TRIAL: NCT05731609
Title: Exploration of the Effectiveness and Feasibility of a Personalized Power Training Program for Youth with Cerebral Palsy Provided Through a Community-tertiary Hospital Partnership
Brief Title: Resistance Intensive Personal Training for Youth with Cerebral Palsy
Acronym: RIPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Elizabeth Condliffe, PhD MD, Clinical Associate Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REB22-1701
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy; Exercise; Resistance Training
Keywords: Cerebral Palsy; CP; Exercise; Strength Training; Power Training; Youth
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Resistance Intensive Personal Training (RIPT) (Experimental): All participants will participate in this arm involving 12 weeks of training 2-3 days/week in a group setting with each session involving 1:1 support for each participant's power training.
  Interventions: Other: Resistance Intensive Personal Training

INTERVENTIONS:
Other: Resistance Intensive Personal Training — Personalized power training program focused on participant goals.

SUMMARY:
Changes related to Cerebral Palsy (CP) include differences in muscle architecture and cortical activity. These result in weakness, decreased functional ability and limited participation in physical activity. Strength training programs, particularly those including power training components, show great potential in improving the gross motor function of youth with CP. However, this intervention is not currently offered in the Calgary area. Delivered via an innovative partnership with community stakeholders, this project will investigate the preliminary effectiveness of the program to enable youth with CP to achieve child and family centered goals. It will also investigate the feasibility of offering this type of program via a community-hospital partnership.

Research Question & Objectives:

1. Can youth with cerebral palsy achieve their goals and improve their motor function through RIPT (Resistance Intensive Personal Training), a power training program offered jointly by specialized physiotherapists and fitness professionals in community settings?
2. What are the barriers and facilitators to delivery of RIPT in a community setting for youth, caregivers, clinicians, and program staff?

DETAILED DESCRIPTION:
Changes related to Cerebral Palsy (CP) include differences in muscle architecture and cortical activity. These result in weakness, decreased functional ability and limited participation in physical activity. Strength training programs, particularly those including power training components, show great potential in improving the gross motor function of youth with CP. However, this intervention is not currently offered in the Calgary area. Delivered via an innovative partnership with community stakeholders, this project will investigate the preliminary effectiveness of the program to enable youth with CP to achieve child and family centered goals. It will also investigate the feasibility of offering this type of program via a community-hospital partnership.

Research Question & Objectives:

1. Can youth with cerebral palsy achieve their goals and improve their motor function through RIPT (Resistance Intensive Personal Training), a power training program offered jointly by specialized physiotherapists and fitness professionals in community settings?
2. What are the barriers and facilitators to delivery of RIPT in a community setting for youth, caregivers, clinicians, and program staff?

Methods:

Study investigators will conduct a mixed-methods experimental prospective cohort study. Two 12-week sessions of RIPT will be offered at the Mount Royal University community recreation centre and delivered in partnership by physiotherapists from Alberta Children's Hospital and community-based fitness professionals with additional support from students at Mount Royal University (training partners). Six youth with CP (aged 8-17, able to follow directions in English and exert a maximal effort with support) will participate in each session with 1:1 support for each participant's power training 1 hour/day, 2-3 days/week in a group setting. At recruitment potential barriers to regular attendance will be explored with an ACH Neurosciences Social Worker available to support as needed. Each participant and their family will generate individual goals using the Canadian Occupational Performance Measure and their individualized program will be tailored to target the movements and muscles needed to achieve each goal by physiotherapists trained in the RIPT protocol.

This study is designed to evaluate if this practical implementation of the program is effective (i.e. can produce similar effect size as measured in randomized-controlled efficacy trials). Motor function will be measured with the gold-standard clinical scale in this population, Gross Motor Function Measure, and objective evaluation of muscle power using the isotonic mode on our Biodex Dynamometer. Both of these outcomes have established effect sizes. Further, study investigators will move the assessment approach to focus on the individual goals identified by the COPM as part of creating the training program by linking each one to the Goal Attainment Scale. For example, a participant's goal to be able to walk to the bus faster, can be objectively evaluated using a validated measure such as the 6-minute Walk Test. Changes in each of these objective outcomes can be prospectively mapped to the Goal Attainment Scale's ordinal rankings to enable repeated-measures analysis of outcomes based on those most salient to an individual. Study investigators will also use EQ-5DY to evaluate quality of life as comments from our pilot clinical program suggest the benefits were quite broad. These outcomes will be collected at baseline 8, and 12 weeks. The change between baseline and 12-weeks represents the key outcome to demonstrate effectiveness. Patient partners feel a shorter program would be more feasible for more participants and one previous study has shown efficacy at 8 weeks. Therefore, the 8-week time point will allow study investigators to explore if participant goals can be met on this shorter timeline.

Following training, youth and their families will complete the Measure of Processes of Care (MPOC 20) and participate in individual family focus-groups. Training partners will complete the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) which are valid and reliable measures of implementation outcomes. Study investigators will also explore the barriers and facilitators to program delivery via semi-structured interviews with the training partners. Interviews will be anonymized and transcribed. Thematic analysis of the transcripts will assess each domain: barriers, facilitators, and perceived impacts of RIPT.

ELIGIBILITY:
Inclusion Criteria:

* At least 8 years old
* 17 years old or younger
* able to follow directions in English
* able to exert maximum effort

Exclusion Criteria:

* Less than 8 years old
* 18 years old or older
* unable to follow directions in English
* unable to exert maximum effort
* acute pathology of the body part to be trained (e.g. injury or surgery)
* A very high degree of neuromotor impairment (GMFCS 5, MACS 4/5) as we are unable to provide mechanical lifts and transfers

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | 14 weeks (from time of consent to end of trial).
  Evidence based outcome measure designed to capture clients self-perception of performance in everyday living over time. Scores are rated on a scale of 1-10, where 1 is the least satisfaction and 10 is the most satisfaction.
Goal Attainment Scale | 14 weeks (from time of consent to end of trial).
  Individualized outcome measure involving goal selection and goal scaling that is standardized in order to calculate the extent to which a patient's goals are met. Scoring is on a scale of -2 to +2, where -2 is no change, 0 is achieving the goal, and +2 is exceeding the goal.

SECONDARY OUTCOMES:
Gross Motor Function Measure | 14 weeks (from time of consent to end of trial).
  Evaluates change that occurs over time in the gross motor function of children with cerebral palsy.
Muscle power assessment | 14 weeks (from time of consent to end of trial).
  Objective measure of muscle power using voluntary contractions based on muscles involved in goal setting for individual participants.
EQ-5D-Y | 14 weeks (from time of consent to end of trial).
  Measure of health related quality of life in children and adolescents. Health is rated on a scale of 1 to 100, where 1 is the worst health and 100 is the best health.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Condliffe, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
There is an open science plan to share de-identified IPD. All data collected in the study will be de-identified and added to a database. Access by other researchers must be requested and agree to a Terms of Use agreement before access is granted.
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available at the end of the study. There is no plan to close the database.
Access Criteria: Researchers requesting access to the database will be required to sign a Terms of Use agreement.